CLINICAL TRIAL: NCT05808517
Title: An Integration of Tai Chi (TC) and Repetitive Transcranial Magnetic Stimulation (rTMS) for Sleep Disturbance in Older Adults
Brief Title: An Integration of Tai Chi and Repetitive Transcranial Magnetic Stimulation for Sleep Disturbance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V1
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Tai Ji; Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TC plus rTMS group (Experimental): Participants received 12 one-hour sessions over 4 weeks (three times per week with a day between sessions). Each session of rTMS consisted of a sequence of three stimulation pulses per string with a string interval of 1 s (total 500 strings, total 1,500 stimulation pulses, and total stimulation time of 30 mins per session). After subjects finished each rTMS session, they immediately attended the TC class together with the participants in the TC-alone group.
  Interventions: Behavioral: Tai Chi; Other: repetitive transcranial magnetic stimulation
- TC-alone group (Active Comparator): Participants underwent a 4-week intervention program consisting of simplified Yang style 12-Form Easy TC given as 1-hour sessions, three times per week. Each session included 5 to 10 minutes of warm-up exercise, 45 minutes of TC practice, and 5 to 10 minutes of cool-down exercise. The TC intervention was conducted in a small group format (i.e., 6-8) led by a trained TC instructor.
  Interventions: Behavioral: Tai Chi
- Treat-as-usual control group (No Intervention): Participants in the TAU control group received treatments as usual for 4 weeks. No additional sleep intervention was provided. All participants were required to complete the subjective and objective assessments.

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi (TC) is a traditional Chinese exercise, also known as a mind-body exercise. It is suitable as an alternative or supplementary form of routine physical exercise for older adults. TC focuses on gentle and rhythmical movements while maintaining a meditative state. Low to moderate activities have benefits to improve sleep disturbances in older adults. In addition, growing evidence widely supports meditation as a potential intervention to improve sleep disturbances through reducing repetitive negative thoughts such as worry and rumination.
  Other Names: TC
  Arms: TC plus rTMS group; TC-alone group
Other: repetitive transcranial magnetic stimulation — The brain stimulation technique repetitive transcranial magnetic stimulation (rTMS) provides the opportunity to non-invasively modulate cortical excitability. In general, low-frequency rTMS (≤ 1 Hz) is thought to inhibit cortical excitability.
  Other Names: rTMS
  Arms: TC plus rTMS group

SUMMARY:
The investigators designed an RCT aimed at 1) exploring the effectiveness of combining TC with rTMS for synergistically improving sleep disturbances in community-dwelling older adults, 2) investigating the mediating roles of arousal states as the underlying mechanism of the potential beneficial effects, and 3) evaluating the feasibility and safety to inform the clinical practice. The investigators hypothesized that integrating TC and rTMS can affect the different dimensions of the arousal system to improve sleep disturbances with optimized clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Classified with sleep disturbances (indications of poor sleep quality with a score >5 in Pittsburgh Sleep Quality Index)
2. Education level at primary or higher, and able to communicate in Cantonese (3) No experience of mind-body exercising such as TC, Qigong, or yoga within the past 6 months

Exclusion Criteria:

1. Serious visual or hearing difficulty
2. Active suicidal ideation or self-harm behaviors
3. Cognitive impairment (a score <26 in the Montreal Cognitive Assessment)
4. Comorbid diagnoses such as mental disorders, organic brain syndrome, or intellectual disabilities
5. Cardiac pacemaker, implanted medication pump, the intracranial implant (e.g., aneurism clips, shunts, stimulators, cochlear implants, or electrodes), or any other metal object within or near the head
6. Receiving other treatments or participating in other clinical trials during the same period
7. Current severe medical condition preventing physical exercise

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The change from baseline (T0) Insomnia Severity Index at immediately after the intervention (T1) and 3-month follow-up (T2) | Baseline (T0), immediately after the intervention (T1), and 3-month follow-up (T2)

SECONDARY OUTCOMES:
The change from baseline (T0) somatic and cognitive arousal assessed by Pre-Sleep Arousal Scale at immediately after the intervention (T1) and 3-month follow-up (T2) | Baseline (T0), immediately after the intervention (T1), and 3-month follow-up (T2)
The change from baseline (T0) cortical arousal measured by 15 minutes eye-closed state electroencephalogram (EEG) at immediately after the intervention (T1) and 3-month follow-up (T2) | Baseline (T0), immediately after the intervention (T1), and 3-month follow-up (T2)
The change from baseline (T0) sleep pattern assessed by an objective measurement (wrist ActiGraph GT3X) at immediately after the intervention (T1) and 3-month follow-up (T2) | Baseline (T0), immediately after the intervention (T1), and 3-month follow-up (T2)
The change from baseline (T0) mood states assessed by Depression, Anxiety, and Stress Scale-21at immediately after the intervention (T1) and 3-month follow-up (T2) | Baseline (T0), immediately after the intervention (T1), and 3-month follow-up (T2)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechinic University, Hong Kong, Hong Kong